CLINICAL TRIAL: NCT06050824
Title: A Comparative Study Between Concomitant Versus Load Therapy in Eradication of Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Hala Hany Shehata, Principle Investigator, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDM0003
Record Dates: First submitted 2023-09-16; First posted 2023-09-22 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concomitant (Active Comparator): Clarithro -pantoprazole- Metronidazole - Amoxicyllin
  Interventions: Drug: Comparing Load and Concomitant therapy
- LOAD (Active Comparator): Levofloxacin -omeprazole- nitazoxanide- Doxycycline
  Interventions: Drug: Comparing Load and Concomitant therapy

INTERVENTIONS:
Drug: Comparing Load and Concomitant therapy — Levofloxacin - Omeprazole - nitazoxanide - doxycycline
  Other Names: Clarithromycin - pantoprazole - Metronidazole - Amoxycyllin

SUMMARY:
All patients who presented with epigastric pain and dyspeptic symptoms will undergo endoscopic gastric biopsies.

The patients will be subjected to: Full history taking, clinical examination, liver function tests, renal function tests, CBC, INR, abdominal ultrasonography.

About 200 patients diagnosed to have H. pylori by infection by microscopically examined, endoscopic gastric biopsies will be enrolled in our study.

All available formalin fixed and paraffin embedded tissue blocks of gastric endoscopic biopsies will be resectioned and stained with Haematoxylin and Eosin. Modified Giemsa stain, and Alcian blue/ PAS stain will be used for verification of Helicobacter pylori and demonstration of intestinal metaplasia respectively.

Biopsies will be classified using the Updated Sydney system of classification of gastritis

DETAILED DESCRIPTION:
The patients will be randomized (closed envelopes) into one of two groups:

1. patients will receive concomitant therapy comprising of pantoprazole (40 mg twice daily), amoxicillin (1 gm twice a day), clarithromycin (500 mg twice a day) and metronidazole (500 mg twice a day) for 2 weeks.
2. patients will receive LOAD therapy comprising of levofloxacin (250 mg with breakfast), omeprazole (40 mg before breakfast), nitazoxanide (Alina) (500 mg twice daily with meals) and doxycycline (100 mg at dinner) for 10 days.

H. Pylori eradication will be confirmed by H. Pylori stool antigen testing at least 4 weeks after cessation of antibiotic therapy with stoppage of PPI therapy at least one to two weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients who presented with epigastric pain and dyspeptic symptoms

Exclusion Criteria:

1. Patients recently (within 6 months) treated with anti-H. pylori therapy.
2. Allergy to any drugs used in our protocol
3. Patients on PPI, antibiotics, and steroid or non-steroidal anti-inflammatory drugs within past one month before randomization.
4. Concomitant significant comorbidities (advanced cardiac, renal, hepatic disease).
5. Presence of GI malignancy.
6. Pregnancy or lactating women.
7. Unable or refuse to give consent. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Eradication of H. pylori infection after treatment | 4 weeks after end of treatment
  Negative stool antigen test for H.pylori

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Helwan University, Cairo, Egypt